CLINICAL TRIAL: NCT03109470
Title: The Durability of Early RA Disease Control After Tocilizumab Withdrawal: A Canadian Experience
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient enrollment potential
Sponsor: Pope Research Corporation (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: PRC-03-2012
Record Dates: First submitted 2013-11-13; First posted 2017-04-12 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Tocilizumab; Early Rheumatoid Arthritis; Observational; Canadian
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who participated in the FUNCTION Study (Protocol WA19926) will be enrolled in this study. The investigators want to learn how long it takes Early Rheumatoid Arthritis patients who were treated with Tocilizumab to require treatment with another biologic medication.

ELIGIBILITY:
Inclusion Criteria:

* Completed 2 years in the FUNCTION (WA19926) trial
* Patient has provided written informed consent and is willing to comply with the requirements of this study protocol

Exclusion Criteria:

* Requirement for immediate treatment with a biologic therapy following completion of the FUNCTION (WA19926) trial as per treating physician judgement.
* Presence of any condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients withdrawing first-line tocilizumab and/or methotrexate therapy due to therapeutic response during the FUNCTION (WA19926) study that have agreed to provide informed consent will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rate of Biologic Treatment | 2 years
  To describe the rate of requiring biologic treatment over 2 years following completion of the FUNCTION study

SECONDARY OUTCOMES:
Treatment after completion of FUNCTION study | Baseline
  To determine the type of RA treatment regimen used by the treating physician upon completion of the FUNCTION study
Rate of requiring treatment intensification | 2 years
  To determine the rate of requiring treatment intensification with a traditional DMARD(s) completion of the FUNCTION study. The durability of response after completion of the FUNCTION study. The clinical measures of disease progression over 2 years after completion of the FUNCTION study. The clinical measures of disease progression over 2 years after completion of the FUNCTION study.
Change in functional status | 2 years
  The change in patient-reported functional status over 2 years after tocilizumab withdrawal or maintaining Mtx or changing DMARD(s)
Work productivity | 2 years
  To determine work productivity over 2 years after completion of the FUNCTION study
Healthcare Utilization | 2 years
  To determine health-care utilization over 2 years after completion of the FUNCTION study

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD, MPH, FRCPC, Principal Investigator — Pope Research Corp.; John S Sampalis, BSc, BA, MSc, PHD, FACE, Principal Investigator — JSS Medical Research Inc.